CLINICAL TRIAL: NCT01509651
Title: Reversal of Rocuronium-induced Neuromuscular Block With Sugammadex in Heart Failure Patients
Brief Title: Sugammadex and Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Guy CAMMU, MD, PhD, Staff Anesthesiologist, Onze Lieve Vrouw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B126201112363
Record Dates: First submitted 2012-01-01; First posted 2012-01-13 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Postoperative Neuromuscular Block
Keywords: antagonists neuromuscular block; neuromuscular block, monitoring; neuromuscular function
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sugammadex (Experimental)
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — After the induction of anaesthesia, monitoring neuromuscular function is initiated and performed continuously using the TOF-Watch SX (Organon Ireland Ltd, Ireland) at the thumb. Repetitive train-of four (TOF) stimulation is applied every 15 s at the ulnar nerve until the end of anaesthesia, at least until recovery of the TOF ratio to 0.9 after administration of sugammadex. Each patient receives a single IV bolus dose of rocuronium 0.6 mg kg-1, after which tracheal intubation is performed. Maintenance doses of rocuronium 0.1 mg kg-1, are permitted as required and administered at the reappearance of the second twitch in the TOF. On reappearance of the second twitch at the end of surgery, patients receive a single IV bolus dose of sugammadex, 2.0 mg kg-1, for reversal.

SUMMARY:
Although anticholinesterase reversal agents have been used in combination with anticholinergic drugs for over half a century, it has been suggested that they should be used with caution in patients with underlying cardiovascular disease. As sugammadex has no endogenous targets, it is unlikely to cause any adverse cardiovascular effects. This selective relaxant binding agent is specifically designed to encapsulate rocuronium, which can, therefore, promptly restore neuromuscular function regardless of any levels of NMB as the dose is increased.

Some reports, however, suggest that sugammadex may have increased time to effect in some patient populations like the elderly, patients in intensive care and renal failure patients. A less dynamic circulation and increased transfer time to the effector site in these subjects are likely explanations for this effect. The present trial was designed to assess the safety and efficacy of sugammadex 2.0 mg kg-1 for the reversal of rocuronium-induced NMB in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 yr or older
* categorized as American Society of Anesthesiologists class 3-4 and New York Heart Association class 2-4
* with an ejection fraction <25%
* scheduled to undergo elective surgery for cardiac resynchronization therapy, an automated implantable cardioverter-defibrillator (ICD), or battery replacement of an ICD or biventricular pacemaker, during general anaesthesia.

Exclusion Criteria:

* expected to have a difficult intubation for anatomic reasons
* they had a neuromuscular disorder
* a personal or family history of malignant hyperthermia
* or known allergy to medication used during general anaesthesia
* not able or willing to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The time from start of sugammadex administration to recovery of the train-of-four (TOF) ratio to 0.9. | Participants will be followed for the duration of recovery from neuromuscular block, an expected average of 10min

SECONDARY OUTCOMES:
The time from start of sugammadex administration to recovery of the TOF ratio to 0.7 and 0.8. | Participants will be followed for the duration of recovery from neuromuscular block, an expected average of 10min
Adverse hemodynamic events. | From anesthesia induction until 3h after arrival in the postanaesthesia care unit (PACU).
Adverse respiratory events (SpO2 <90% and/or signs of airway obstruction). | From arrival in the PACU until 30min thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Cammu, MD, PhD, Principal Investigator — OLV Hospital, Anesthesiology and CCM, Aalst, Belgium
Locations (1):
- OLV Hospital, Aalst, Belgium

REFERENCES:
- [Background] Sorgenfrei IF, Norrild K, Larsen PB, Stensballe J, Ostergaard D, Prins ME, Viby-Mogensen J. Reversal of rocuronium-induced neuromuscular block by the selective relaxant binding agent sugammadex: a dose-finding and safety study. Anesthesiology. 2006 Apr;104(4):667-74. doi: 10.1097/00000542-200604000-00009. PMID 16571960
- [Background] Dahl V, Pendeville PE, Hollmann MW, Heier T, Abels EA, Blobner M. Safety and efficacy of sugammadex for the reversal of rocuronium-induced neuromuscular blockade in cardiac patients undergoing noncardiac surgery. Eur J Anaesthesiol. 2009 Oct;26(10):874-84. doi: 10.1097/EJA.0b013e32832c605b. PMID 19455040
- [Background] Suzuki T, Kitajima O, Ueda K, Kondo Y, Kato J, Ogawa S. Reversibility of rocuronium-induced profound neuromuscular block with sugammadex in younger and older patients. Br J Anaesth. 2011 Jun;106(6):823-6. doi: 10.1093/bja/aer098. Epub 2011 Apr 29. PMID 21531745
- [Background] Staals LM, Snoeck MM, Driessen JJ, Flockton EA, Heeringa M, Hunter JM. Multicentre, parallel-group, comparative trial evaluating the efficacy and safety of sugammadex in patients with end-stage renal failure or normal renal function. Br J Anaesth. 2008 Oct;101(4):492-7. doi: 10.1093/bja/aen216. Epub 2008 Jul 23. PMID 18653492